CLINICAL TRIAL: NCT00861978
Title: St. John's Wort Extract LI 160 for the Treatment of Atypical Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cassella-med GmbH & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160DE0838A
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Atypical Depression
Keywords: mild to moderate depression with atypical features according to DSM-IV
MeSH Terms: interventions — Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: St. John's Wort extract

INTERVENTIONS:
Drug: St. John's Wort extract — Coated tablets (batch no. 02080277) containing 300 mg of St. John's Wort extract LI 160 (drug-extract ratio 3-6:1; extraction solvent: 80% Methanol in water; batch no. 02019073) administered orally twice daily (morning and evening) with some liquid for 8 weeks
  Other Names: Jarsin; LI 160
  Arms: 2
Drug: Placebo — Coated placebo tablets (batch no. 01010177) that were identical in shape, size, taste and color were administered orally twice daily (morning and evening) with some liquid for 8 weeks.
  Arms: 1

SUMMARY:
The aim of tis study is to assess the efficacy and safety of Jarsin® 300 mg as an acute treatment in mild to moderate depression with atypical features.

DETAILED DESCRIPTION:
The general picture of depression is still that of the traditionally called endogenous type, which is also the form that was characterized extensively in clinical trials. Atypical depression with reversed vegetative signs, such as hyperphagia or hypersomnia, is traditionalla neglected, demonstrated by the fact that in the most widely used depression scales, such as the Hamilton Depression Scale, melancholic symptoms have a specific weight, while, by contrast, reversed vegetative signs are not included. This etablishes a tendency to underestimate the severity of atypical depression.

ELIGIBILITY:
Main Inclusion Criteria:

* Mild to moderate depression (ICD-10 F32.0, F32.1) with atypical features according to DSM-IV, lasting at least 3 months
* Female and male Caucasians aged 18 to 70 years
* At least one of HAMD-28 scale items 22-26 scores >1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2002-12; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)